CLINICAL TRIAL: NCT04107792
Title: The Impact of an Education Workshop on Parental Sense of Competence
Brief Title: Parental Sense of Competence Workshops for Parents of Children With Sensory Processing Issues
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Yani Hamdani, PhD, Adjunct Scientist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPIStudy
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Parents
Keywords: parenting; parental sense of competence; children; sensory processing issues

STUDY DESIGN:
Intervention Model Description: pilot randomized waitlist control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Parents of children with sensory processing issues who attend Workshop 1
  Interventions: Behavioral: parental sense of competence workshop
- Waitlist Control (No Intervention): parents of children with sensory processing issues who attend Workshop 2

INTERVENTIONS:
Behavioral: parental sense of competence workshop — The intervention will be a two-hour parent education workshop that provides education and teaches parent-mediated strategies for managing children's behaviours associated with SPIs.
  Arms: Experimental

SUMMARY:
The primary objective of this pilot randomized waitlist control trial is to evaluate the impact of an OT-led parent education workshop on the PSOC of parents of children experiencing SPIs who are on the waitlist for a neurodevelopmental diagnostic assessment. The secondary objective is to obtain a subjective evaluation of the content, format, and delivery of the parent education workshop from the parents' perspectives.

DETAILED DESCRIPTION:
Introduction. Parents of children with sensory processing issues (SPIs) experience decreased levels of parental sense of competence (PSOC) in managing SPI-related behaviours that challenge conventional parenting skills. Occupational therapy (OT)-led parent education workshops (PEWs) have been found to increase the PSOC of parents of children with SPIs who have a formal Autism Spectrum Disorder (ASD) diagnosis. However, research is limited on how these interventions affect PSOC of parents of children with SPIs who do not have a formal diagnosis, and are still on the waitlist for a neurodevelopmental assessment. This is vital as children with SPIs and their parents may have limited access to specialist referrals, government-funded interventions, or support services while they await a diagnostic assessment. SPI-related workshops may provide an opportunity to support families and promote PSOC and well-being by providing strategies to address SPI-related behaviours while they wait (which may be beneficial regardless of whether their child eventually receives a formal neurodevelopmental diagnosis or not). Objectives. The primary objective of this pilot randomized waitlist control trial is to evaluate the impact of an OT-led parent education workshop on the PSOC of parents of children experiencing SPIs who are on the waitlist for a neurodevelopmental diagnostic assessment. The secondary objective is to obtain a subjective evaluation of the content, format, and delivery of the parent education workshop from the parents' perspectives. Methods. Parents will be recruited from the waitlist for a neurodevelopmental assessment for their children through the "Communication, Learning, and Behaviour" clinic at Holland Bloorview Kids Rehabilitation Hospital. Participants will be randomly selected to attend one of two identical workshops scheduled two weeks apart. The PSOC Scale, along with demographics and follow-up questionnaires that include both closed and open-ended questions, will be administered to parents pre- and post-workshop attendance. Descriptive statistics, an independent sample t-test and a two-way Analysis of Variance (ANOVA) will be used to analyze quantitative data from these outcome measures. To analyze the qualitative data (parents' open ended responses on the follow-up feedback questionnaire), a content analysis will be completed, which will be used to complement the quantitative results, as well as provide feedback regarding the content, format, and delivery of the parent education workshop. Practice Implications. Results from this study can provide evidence to support the need for parent education workshops in improving the PSOC of parents of children on the waitlist for a neurodevelopmental assessment, promote mental health and wellbeing of parents while they wait for the assessment, promote parenting that helps children with SPIs engage in daily life occupations, and inform the development of future workshops. Conclusion. Information garnered from this study can inform the development of OT services that can address the current gap in care while parents and their children with SPIs are waiting for a formal neurodevelopmental assessment and referrals to publicly funded services funded for specific diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with Sensory Processing Issues
* On the waitlist for a neurodevelopmental diagnostic assessment at the "Communication, Learning, and Behaviour" clinic at Holland Bloorview Kids Rehabilitation Hospital
* At least 18 years of age or older
* Target child(ren) with SPIs must be between the ages of 0-17 years (which is the age restriction of the Parental Sense of Comptence scale)
* The child(ren)'s scheduled neurodevelopmental diagnostic assessment date must be after their final completion of the Parental Sense of Competence Scale (two weeks following workshop attendance) to control for any external influence that a formal diagnosis may have on participants' Parental Sense of Competence
* Basic English comprehension reading and writing skills
* Access to the internet

Exclusion Criteria:

* Previously attended a parent education workshop or intervention targeting Sensory Processing Issues
* Attend a different parent education workshop or intervention for Sensory Processing Issues throughout the duration of the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Parental Sense of Competence (PSOC) Scale | One Month
  The Parental Sense of Competence (PSOC) scale is a self-report scale that measures and assesses parent self-efficacy on two dimensions: Satisfaction and Self-Efficacy. It is a 17-item scale, with each item rated on a 6-point Likert scale, anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". Nine (9) items (#2, 3, 4, 5, 8, 9, 12, 14, 16) on the PSOC are reverse coded. Once reverse coded, the score for each item is added up to give the "total score" for this scale. The minimum and maximum total scores (total range) are 17 and 102, respectively. No subscale scores are reported. A higher total score indicates a higher parenting sense of competency; a lower total score indicates a lower parenting sense of competency. There are no average scores or "cut offs" for this tool.

CONTACTS AND LOCATIONS:
Overall Officials: Yani Hamdani, PhD, Principal Investigator — University of Toronto
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No